CLINICAL TRIAL: NCT00973947
Title: A Prospective Randomised Controlled Clinical Trial Investigating the Benefits of Patient-customised Headrests Versus Standard (Non-patient Specific) Headrests in the Immobilisation of Patients Receiving Radiotherapy for Head and Neck Cancer
Brief Title: Customized Headrest or Standard Headrest in Holding Patients Still While Undergoing Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-09 ICORG; ICORG-08-09; EU-20954
Record Dates: First submitted 2009-09-05; First posted 2009-09-09 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2013-01

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; metastatic squamous neck cancer with occult primary squamous cell carcinoma; untreated metastatic squamous neck cancer with occult primary; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent lymphoepithelioma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; recurrent metastatic squamous neck cancer with occult primary; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Radiotherapy, Conformal

ARMS (2):
- Control (Other): Immobilisation: Standard headrest plus individual customised mask (orfit)
  Interventions: Other: questionnaire administration; Radiation: 3-dimensional conformal radiation therapy; Radiation: radiation therapy treatment planning/simulation
- TRial Arm (Other): Immobilisation: Customised headrest plus individual customised mask (orfit)
  Interventions: Other: questionnaire administration; Radiation: 3-dimensional conformal radiation therapy; Radiation: radiation therapy treatment planning/simulation

INTERVENTIONS:
Other: questionnaire administration
Radiation: 3-dimensional conformal radiation therapy
Radiation: radiation therapy treatment planning/simulation

SUMMARY:
RATIONALE: Using a customized headrest to hold patients in one position may help doctors plan treatment for patients with head and neck cancer. It is not yet known whether a customized headrest is more effective than a standard headrest in holding patients still during radiation therapy.

PURPOSE: This randomized clinical trial is studying a customized headrest to see how well it works compared with a standard headrest in holding patients still while undergoing radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate and compare the treatment set-up accuracy of customized vs standard headrest in immobilizing patients undergoing radiotherapy for head and neck cancer.
* To determine and compare patient comfort with the two immobilization techniques.

Secondary

* To evaluate radiation therapists' satisfaction with the two immobilization techniques.
* To examine and compare the cost effectiveness of the two immobilization techniques.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 arms.

* Arm I: Patients are immobilized using the standard thermoplastic four-point fixation mask and the standard headrest system. Patients undergo 3-dimensional conformal radiotherapy as per standard of care.
* Arm II: Patients are immobilized using the standard thermoplastic four-point fixation mask and the customized headrest system. Patients undergo 3-dimensional conformal radiotherapy as per standard of care.

Patients score their comfort using the Visual Analogue Scale during the course of radiotherapy. Radiation therapists complete an evaluation questionnaire for each treatment planning and procedure.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed head and neck malignancy
* Planning to undergo radical 3-dimensional conformal radiotherapy (using the Oncentra MasterPlan treatment planning system) at St Luke's Hospital

PATIENT CHARACTERISTICS:

* No evidence of any other significant clinical disorder or laboratory finding that would make it undesirable for the patient to participate in the study
* Able to comply with the study, in the opinion of the researcher and/or medical team

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Treatment set-up accuracy | 2010
Patient comfort with the two immobilization techniques as assessed by a patient-scored Visual Analogue Scale | 2010

SECONDARY OUTCOMES:
Radiation therapists' satisfaction as assessed by a questionnaire | 2010
Cost-effectiveness as assessed by resource implications of the two immobilization techniques | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Thirion, MD, Principal Investigator — Saint Luke's Hospital
Locations (1):
- Saint Luke's Hospital, Dublin, Ireland